CLINICAL TRIAL: NCT07348289
Title: PIVO-ED: Protocol for Intermountain Venous Access Optimization for Blood Cultures in the Emergency Department
Brief Title: PIVO Use for Blood Cultures in the Emergency Department
Acronym: PIVO-ED
Status: Recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1053426; PIVO-ED (Other: BD)
Record Dates: First submitted 2025-12-11; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Device Performance; Emergency Medicine
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients in whom PIVO is used: This cohort includes patients in whom PIVO is used to assess successful use of the device and contamination rates among blood cultures obtained.
  Interventions: Device: PIVO device, a needle-free blood draw device
- Blood cultures obtained without PIVO use: This comparison group includes patients in whom the PIVO device is not used for comparison to blood cultures in which it is used.

INTERVENTIONS:
Device: PIVO device, a needle-free blood draw device — The PIVO device, a needle-free blood draw device, may be used through an IV to obtain a blood sample and extends beyond the IV to ideally reduce the potential for contamination and to improve success in obtaining a sample.
  Per Google AI: "PIVO™ by Velano Vascular stands for Peripheral IV Origin, a needle-free blood draw device that uses a patient's existing peripheral IV (PIV) line to collect blood, avoiding extra needle sticks and reducing pain, hemolysis, and contamination, facilitating the "One-Stick Hospital Stay" goal for better patient care."
  Groups: Patients in whom PIVO is used

SUMMARY:
The investigators will implement a protocol for use of the PIVO device for blood culture collection in the emergency department. This protocol utilizes the device in various scenarios to reduce needlesticks while allowing for accurate and appropriate assessment of potential pathogens in the bloodstream. The study team will train staff on use of the device then monitor utilization and contamination rates among emergency department patients.

DETAILED DESCRIPTION:
This prospective implementation and efficacy study will be conducted with primary implementation at three Intermountain Health emergency departments: Park City Hospital (Park City, Utah), Primary Children's Hospital (Salt Lake City, Utah), and Utah Valley Hospital (Provo, Utah). These three sites have a combined annual emergency department visit volume exceeding 100,000 visits, ensuring a robust implementation setting for the evaluation of blood culture practices. The investigators will seek to expand the protocol to three secondary sites, pending the results of the initial data regarding blood culture contamination rates from the primary sites. These secondary sites include the emergency departments at Intermountain Medical Center (Murray, Utah). LDS Hospital (Salt Lake City, Utah), and McKay-Dee Hospital (Ogden Utah). These sites have combined annual emergency department volumes exceeding 150,000 patients per year.

The study will launch on October 1, 2025, following the system-wide Epic EHR deployment in September 2025. During October, each ED will undergo a structured training program for clinical staff, including ED nurses, physicians, and phlebotomists. This training will focus on the indications for PIVO use, technical instructions, workflow integration, and documentation standards within Epic. After training, the PIVO protocol will be implemented for a total study duration of 13 months, with data collection occurring between November 2025 and October 2026. The investigators will perform interim analyses at three, six, and nine months to assess PIVO utilization and any need for site-specific re-training, feedback, and intervention. The study team will perform a REDCap-based survey of relevant practitioners (phlebotomists, laboratory technicians, and nurses) who have utilized the device at ten months to assess their comfort with use and willingness to recommend the device. All individuals who have performed at least one blood culture draw utilizing the PIVO will be eligible to participate. The study team will distribute the survey link through site clinical leaders to relevant groups who perform these draws, and they will be asked to participate if they have utilized the PIVO. Investigators will obtain informed consent for participation per Intermountain IRB procedures.

After the review of blood culture results and contamination rates at three months, as well as feedback from the primary site clinical leaders regarding the efficacy and ease of use of the PIVO, the study team will work with clinical leaders at the secondary sites of Intermountain Medical Center, LDS Hospital, and McKay-Dee Hospital to expand the protocol to these emergency departments. Currently, Intermountain Medical Center and LDS Hospital do not utilize the PIVO; the team will provide training and take necessary steps for implementation pending approval from clinical leaders within these sites. McKay-Dee Hospital is currently using the PIVO but will also likely require training specific to its use within this protocol in the emergency department setting. The investigators will aim to have implementation of the protocol within these sites at the six-month mark with ongoing data collection related to blood culture contamination rates across all sites over the entire study period.

Based on historical data and protocol-defined inclusion criteria, the investigators estimate that approximately 5,000 total blood cultures will be collected across the three primary EDs during the one-year study period. Pending adoption of the protocol at the secondary sites, the team would anticipate an additional 5,000 total blood cultures performed in these emergency departments over six months. The investigators anticipate that approximately 40% (4,000 blood cultures) will involve the PIVO device. The remaining 6,000 cultures will be collected via standard venipuncture practices. The investigators expect that for the large majority of the cultures obtained with the PIVO device, patients will have also had a blood culture performed using standard procedures.

The PIVO utilization protocol involves three scenarios. In all three scenarios, blood culture draws using PIVO will occur within 24 hours of IV placement, which is in line with the FDA approval for this indication and per guidance from the manufacturer (BD) regarding this approval.

1. Scenario 1: For patients in whom a second IV is not required, a second blood culture may be obtained using the existing IV with the PIVO device with the condition that this second culture is obtained at least fifteen minutes after the first blood culture. The first blood culture will be obtained using standard procedures at the time of the IV placement. The time of the second culture will be recorded according to current Intermountain procedures.
2. Scenario 2: If a patient already has a peripheral IV in place when blood cultures are ordered, the PIVO device will be used to obtain the first culture through that IV. The second blood culture may be collected through a new stick at a separate site, through the existing IV site using the procedure outlined in scenario 1 (drawn at least fifteen minutes after the first culture), or through a second IV site (if present) using the PIVO device at that site.
3. Scenario 3: For patients in whom a second IV and blood culture from a separate site cannot be obtained within 3 attempts or 5 minutes, the second sample may be collected using the PIVO device through the existing IV site.

To assess clinician satisfaction, a standardized survey tool will be administered to ED staff who use the PIVO device at the study's ten-month mark. The study will utilize the validated System Usability Scale survey with adjustments to reflect use of the PIVO device (see "Clinician Survey"). This tool will include 5-point Likert scale items evaluating: ease of use, comfort using the device, workflow impact, provider assessment of patient comfort, and likelihood of recommending the device to colleagues. The survey will be pilot tested with approximately ten clinicians to assess clarity and usability. Feedback from this pilot will inform revisions prior to wider deployment. For research purposes, all survey responses will be collected anonymously.

To assess contamination rates, all blood cultures will be classified as contaminated or non-contaminated utilizing Intermountain's current review process. For blood cultures classified as contaminated, two study investigators, blinded to collection method, will evaluate each case using Intermountain Health's standard contamination criteria, such as presence of skin flora in a single bottle without clinical indicators of infection. In ambiguous cases, adjudication will be supported by Infectious Disease consultation and reference to peer-reviewed criteria from the literature. In cases of disagreement between reviewers, a third reviewer will resolve the discrepancy.

The study will compare contamination rates in PIVO-collected cultures to those collected via standard methods. The benchmark contamination rate for Intermountain EDs is approximately 1.2%. To evaluate non-inferiority, the study team will use a margin of 0.8%. Based on our expected sample size (4,000 PIVO cultures, 6,000 standard cultures), the investigators estimate the study will have over 80% power to demonstrate that the PIVO group is non-inferior, provided the contamination rate does not exceed 2%. The research team will compare PIVO-related contamination rates to the contamination rates for non-PIVO cultures over the study period at the study sites and will perform a secondary analysis to compare contamination rates by facility.

The study team will perform interim analyses at three, six, and nine months to compare contamination rates between PIVO-obtained cultures and non-PIVO cultures across all included sites. The investigators will present this data to ED medical directors and laboratory leadership to either support the continued use of PIVO in their emergency departments or to discontinue its use (guided by statistical analysis demonstrating evidence of inferiority for blood culture contamination).

Data will be captured via Epic reporting tools, device usage logs, and manually adjudicated culture reviews. Variables will include: demographics (e.g., age, sex), culture method (PIVO vs. standard), success/failure of venipuncture, indication for PIVO use, microbiologic results (including contamination status), results of clinical testing, method and site of obtaining the blood culture, and survey responses from clinicians.

Statistical analysis will include descriptive statistics, proportions with 95% confidence intervals, and comparisons using chi-square or Fisher's exact tests. The study team will perform additional assessment of contamination rates using Newcombe and Miettinen scores with Nurminen confidence intervals around differences, comparing lower bounds to the non-inferiority margin. Subgroup analyses will be conducted by site and provider role. Final analysis and manuscript preparation will occur in October 2026 following full adjudication of all cultures.

ELIGIBILITY:
Inclusion Criteria: Patients in whom blood cultures are obtained in the emergency department.

-

Exclusion Criteria: none

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study evaluates patients in whom blood cultures are obtained in the emergency department during the study period. The primary population of interest is those in whom the PIVO device is used, with comparison to the overall population of patients in whom blood cultures are obtained.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
PIVO utilization | From baseline until 12 months after baseline
  The investigators will assess utilization of the device for blood cultures obtained in the emergency department through review of the medical record and documentation of cases in which PIVO was used for blood cultures as a proportion of all blood cultures obtained.
Contamination rates | From baseline until 12 months after baseline
  The investigators will assess contamination rates for blood cultures obtained using the device compared to blood cultures obtained without the device.

SECONDARY OUTCOMES:
Staff satisfaction and willingness to recommend the device | Six months after study initiation
  The investigators will survey staff who have utilized the PIVO device to assess their satisfaction with use and willingness to recommend this to others.

CONTACTS AND LOCATIONS:
Locations (1):
- Park City Hospital, Park City, Utah, United States

IPD SHARING:
Plan to Share IPD: No